CLINICAL TRIAL: NCT00474812
Title: Phase II Study of Dasatinib (BMS-354825) in Patients With Metastatic Adenocarcinoma of the Pancreas
Brief Title: Dasatinib in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00228; NCI-2009-00228 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000546554; CASE 5206; CASE 5206 (Other: Case Western Reserve University); 7828 (Other: CTEP); U01CA062502 (NIH)
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2013-11

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib Treatment (Experimental): Patients receive oral dasatinib twice daily on days 1-28.
  Interventions: Drug: dasatinib; Procedure: laboratory biomarker analysis; Procedure: physiologic testing

INTERVENTIONS:
Drug: dasatinib
  Other Names: BMS-354825; Sprycel
Procedure: laboratory biomarker analysis — Correlative study
Procedure: physiologic testing — Correlative study
  Other Names: study of physiologic variables

SUMMARY:
Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This phase II trial is studying how well dasatinib works in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the overall survival, including median survival, of patients with metastatic adenocarcinoma of the pancreas treated with dasatinib.

SECONDARY OBJECTIVES:

I. Determine the effects of this drug on quantities of circulating tumor cells in these patients.

II. Determine the time to progression in patients treated with this drug. III. Determine pre- and post-drug fat-free mass and gait speed in patients treated with this drug.

IV. Evaluate the toxicity of this drug in these patients. V. Evaluate objective response rate in patients treated with this drug.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral dasatinib twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection at baseline and during days 25-31. Samples are analyzed for quantification of circulating tumor cells. Patients also undergo analysis of fat-free mass and gait speed at baseline and at 1, 2, and 6 months.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* Metastatic disease
* Measurable or evaluable/nonmeasurable disease
* No known brain metastases
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* Absolute granulocyte count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin > 8.5 g/dL
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* AST and ALT =< 2.5 times ULN
* Creatinine =< 2.0 mg/dL
* Not pregnant or nursing
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to dasatinib
* No QTc prolongation (i.e., QTc interval >= 480 msecs [Fridericia correction]) or other significant ECG abnormalities
* LVEF normal by MUGA scan
* No condition that impairs ability to swallow and retain dasatinib tablets, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* No clinically significant cardiovascular disease, including any of the following:

  * Myocardial infarction or ventricular tachyarrhythmia within the past 6 months
  * Major conduction abnormality (unless a cardiac pacemaker is present)
* Recovered from all prior therapy
* More than 4 weeks since prior adjuvant chemotherapy (6 weeks for nitrosoureas or mitomycin C) and/or radiotherapy
* No prior chemotherapy for metastatic disease
* More than 4 weeks since prior EGFR inhibitors (e.g., imatinib mesylate, gefitinib, erlotinib hydrochloride, or lapatinib ditosylate)
* No prior EGFR inhibitors that target Src kinases
* At least 7 days since prior and no concurrent agents with proarrhythmic potential
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent grapefruit or grapefruit juice
* No other concurrent anticancer agents or therapies
* No concurrent systemic antacids (i.e., H2-receptor antagonists and proton pump inhibitors) [Locally acting antacids (e.g., Maalox, Mylanta) allowed within either 2 hours before or 2 hours after dasatinib therapy]
* No concurrent uncontrolled illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * History of significant bleeding disorder, including congenital (von Willebrand's disease) or acquired (anti-factor VIII antibodies) disorders
  * Large pleural effusions
  * Psychiatric illness or social situation that would preclude study compliance
* More than 7 days since prior and no concurrent CYP3A4 inducers or inhibitors
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-05; Primary Completion 2013-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Nock, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Cleveland, Ohio area hospitals, Case Medical Center University Hospitals and MetroHealth Medical Center.
Period: Overall Study
Arm/Group | Dasatinib Treatment
Started | 51
Completed | 44
Not Completed | 7
Not completed — Withdrawal by Subject | 5
Not completed — No Initiation of treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib Treatment
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 61 [43 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 46
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival
Description: From the date of onset of treatment to the date of death and to the date of last follow-up for those still alive, assessed up to 24 months
Time Frame: assessed up to 24 months
Population: Intent to treat.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib Treatment
Number analyzed (Participants) | 51
months | 4.7 [2.8 to 6.9]

2. Secondary Outcome: Objective Response Rate (Complete Response, Partial Response, or Stable Disease), Evaluated Using the New International Criteria Proposed by the RECIST Committee
Description: Response is defined as CR (Complete Response), PR (Partial Response) or SD (Stable Disease) per Response Evaluation Criteria in Solid Tumor (RECIST criteria). Possible evaluations include: CR: Disappearance of all target lesions. PR: At least a 30% decrease in the size of target lesions. SD: neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as progressive disease (PD). Progressive disease (PD) is defined as: at least a 20% increase in the sum of the LD of target lesions.
Time Frame: Up to 5 years
Population: Patients that reached first scans at 2 months
Measure: Number; unit: participants
Arm/Group | Dasatinib Treatment
Number analyzed (Participants) | 34
participants
  Progressive disease | 24
  Stable Disease | 10

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Number of months patients were free of disease progression, defined as < 20% increase in the sum of the LD of target lesions nor the appearance of one or more new lesions.
Time Frame: Up to 5 years
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib Treatment
Number analyzed (Participants) | 51
months | 2.1 [1.6 to 3.2]

4. Secondary Outcome: Gait Speed
Description: Gait speed, determined by a 4 meter walk along a properly measured stretch of hallway while being timed with a stopwatch.
Time Frame: baseline
Population: Participants who were ambulatory at baseline
Measure: Mean (Standard Error); unit: meters per second
Arm/Group | Dasatinib Treatment
Number analyzed (Participants) | 17
meters per second | 4.1 (0.32)

5. Secondary Outcome: Gait Speed
Description: as for outcome 4
Time Frame: at 8 weeks
Population: Participants who were ambulatory at 8 weeks
Measure: Mean (Standard Error); unit: meters per second
Arm/Group | Dasatinib Treatment
Number analyzed (Participants) | 10
meters per second | 4.6 (0.64)

ADVERSE EVENTS:
Time Frame: Adverse Events that occur during treatment or within 30 Days of the last dose. The time frames for patients was 0-23 months.
Arm/Group | Dasatinib Treatment
Serious Adverse Events (participants affected / at risk) | 21/51
Other Adverse Events (participants affected / at risk) | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib Treatment (N=51)
Abdominal pain (Gastrointestinal disorders) | 2
Cardiac Troponin Increase (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Death not associated with CTCAE term - Death NOS (not otherwise specified) (General disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Hepatobiliary disorders (Hepatobiliary disorders) | 2 — Increased liver function tests
Hepatobiliary disorders (Hepatobiliary disorders) | 1 — cholangitis
Infections and infestations - Other, NOS (Infections and infestations) | 8
Myocardial Infarction (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Nervous system disorders - Other, NOS (Nervous system disorders) | 1
Pain (General disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 2
Sinus bradycardia (Cardiac disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Thromboembolic event (Vascular disorders) | 5
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib Treatment (N=51)
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 34
Agitation (Psychiatric disorders) | 3
Alanine aminotransferase increased (Investigations) | 27
Alkaline phosphatase increased (Investigations) | 34
Alopecia (Skin and subcutaneous tissue disorders) | 4
Anemia (Blood and lymphatic system disorders) | 36
Anorexia (Metabolism and nutrition disorders) | 34
Anxiety (Psychiatric disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Aspartate aminotransferase increased (Investigations) | 35
Back pain (Musculoskeletal and connective tissue disorders) | 13
Blood bilirubin increased (Investigations) | 11
Chills (General disorders) | 8
Confusion (Psychiatric disorders) | 4
Constipation (Gastrointestinal disorders) | 23
Creatinine increased (Investigations) | 7
Dehydration (Metabolism and nutrition disorders) | 15
Depression (Psychiatric disorders) | 11
Diarrhea (Gastrointestinal disorders) | 20
Dizziness (Nervous system disorders) | 8
Dry mouth (Gastrointestinal disorders) | 4
Dysgeusia (Nervous system disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Edema face (General disorders) | 9
Edema limbs (General disorders) | 8
Fatigue (General disorders) | 39
Fever (General disorders) | 8
Gastrointestinal disorders - Other, NOS (Gastrointestinal disorders) | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 12
Headache (Nervous system disorders) | 8
Hot flashes (Vascular disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 26
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypertension (Vascular disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 31
Hypocalcemia (Metabolism and nutrition disorders) | 25
Hypoglycemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 18
Hyponatremia (Metabolism and nutrition disorders) | 31
Hypophosphatemia (Metabolism and nutrition disorders) | 7
INR increased (Investigations) | 3
Insomnia (Psychiatric disorders) | 18
Lymphocyte count decreased (Investigations) | 26
Mucositis oral (Gastrointestinal disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 33
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 10
Platelet count decreased (Investigations) | 16
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11
Thromboembolic event (Vascular disorders) | 3
Vomiting (Gastrointestinal disorders) | 25
Weight loss (Investigations) | 18
White blood cell decreased (Investigations) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less